CLINICAL TRIAL: NCT01847196
Title: A Multi-center, Early Feasibility Study of the Angel® Catheter in Critically Ill Subjects at High Risk of Pulmonary Embolism
Brief Title: Angel® Catheter Early Feasibility Clinical Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IDE approval received for larger Pivotal Study
Sponsor: BiO2 Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QD-155
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis; Venous Thromboembolism
Keywords: Pulmonary Embolism; PE; DVT; Deep Vein Thrombosis; VTE; Venous Thromboembolism; prophylaxis; thromboprophylaxis; contraindications to thromboprophylaxis; prophylactic; prevention; Inferior vena cava filter; IVC filter; filter; prevention of pulmonary embolism; trauma; critically-ill
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis; Venous Thromboembolism; Wounds and Injuries; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Angel® Catheter (Experimental): All eligible subjects will receive an Angel® Catheter.
  Interventions: Device: Angel® Catheter

INTERVENTIONS:
Device: Angel® Catheter — The Angel® Catheter combines the functions of an inferior vena cava (IVC) filter and a multi-lumen central venous catheter (CVC). The device is designed to be placed in the inferior vena cava, via the femoral vein, for the prevention of Pulmonary Embolism (PE), and for access to the central venous system. The device is intended for short-term use (less than 30 days) and must be removed before hospital discharge.
  Other Names: Angel Catheter; 2011-0420

SUMMARY:
The primary objective of this clinical trial is to obtain initial insights into the safety of the Angel® Catheter in critically ill subjects with high risk of venous thromboembolism (VTE) disease AND who are not receiving pharmacological thromboprophylaxis.

DETAILED DESCRIPTION:
STUDY ENDPOINTS

1. Primary Endpoints:

   a. Initial Insights into Safety
   * Success in delivery, maintenance and removal of the Angel® Catheter.
   * Incidence and seriousness of all adverse events.
   * Incidence of device or procedure-related adverse events.
2. Secondary Endpoints:

   * Evaluation of the separate and combined functions of the IVC filter and the central venous catheter device.
   * Evaluate investigative site's ability to comprehend the procedural steps (Per the Insertion Procedure, the Repositioning Procedure, and the Removal Procedure)
   * Evaluate operator challenges with device use (human factors).
   * Evaluate success and challenges encountered in conducting a pivotal trial in critically ill patient population - including but not limited to Informed Consent and enrollment.

ENROLLMENT AND SUBJECT SAMPLE SIZE

The study is expected to enroll up to 20 subjects in up to 4 US investigational sites with a goal for 10 evaluable subjects in whom Angel® Catheter placement has been attempted.

STUDY DURATION

The device is designed to be deployed for less than 30 days. After enrollment and Angel® Catheter placement, subjects will be followed daily through the post-removal, seven (7) day follow up or until hospital discharge, whichever occurs first.

ELIGIBILITY:
INCLUSION CRITERIA (Must Answer YES to all Inclusion Criteria):

1. Subject or legally authorized representative is willing and able to provide written informed consent, AND
2. Subject is 18 years or older, AND
3. Subject is currently admitted OR to be admitted to the Intensive Care Unit (ICU) within ≤36 hours of screening, AND
4. Subject has a clinical need for a Central Venous Catheter, and/or the subject has an existing Central Venous Catheter that has been in place for <36 hours before Angel® Catheter placement, AND
5. Subject is considered at high risk for PE and meets ONE of the following criteria:

   1. Subject has multiple trauma with at least ONE of the following:

      * Severe head injury
      * Head injury with a long bone fracture
      * Spinal cord injury with paraplegia or quadriplegia
      * Multiple (≥2) long bone fractures
      * Multiple (≥2) long bone fractures with pelvic fracture
      * Pelvic fracture requiring open fixation
   2. Critically ill subject in the Intensive Care Unit with at least ONE of the following:

      * Hemorrhagic or ischemic stroke
      * Multiple organ failure
      * Active or recent bleeding (within the past 2 weeks)
      * Severe sepsis
      * Lower extremity DVT
      * Anticipated ventilator requirement of greater than one week
   3. Critically ill subject requiring temporary (≥48 hours) interruption of medical thromboprophylaxis (prophylactic anticoagulation)

EXCLUSION CRITERIA (Must Answer NO to All Exclusion Criteria):

1. Subject is pregnant or lactating
2. BMI = (Weight (lb) x 703)/(〖Height〗^2 (inches)) > 45; BMI may also be calculated at http://nhlbisupport.com/bmi/bminojs.htm
3. Subject has a pre-existing IVC filter in place
4. Subject is currently receiving prophylactic anticoagulation, other than aspirin or Plavix. Specifically, the subject is receiving any of the following medications: heparin, low molecular weight heparin, factor Xa inhibitors (i.e. xabans), Coumadin, and thrombin inhibitors.
5. Subject has a diagnosis of pulmonary embolism
6. Subject is participating in another clinical investigation
7. Subject has known hypersensitivity to any of the components of the Angel® Catheter, specifically Nitinol (nickel and/or titanium)
8. Subject has functioning pelvic renal allograft on the only side available for device insertion
9. Subject has undergone a surgical procedure involving the femoral vein or pelvic veins through which the device must be inserted
10. Anatomic inability to place the Angel® Catheter (including a history of thrombosis of venous system on side of proposed access)
11. Anticipated survival ≤48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schreiber, MD, Principal Investigator — Oregon Health and Science University; Larry Martin, MD, Principal Investigator — University of Mississippi Medical Center; John Holcomb, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Michael Cripps, MD, Principal Investigator — University of Texas Southwestern Medical Center (Dallas)
Locations (4):
- United States (4):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For this study, enrollment was defined as the time of consent. There was a possibility that a consented subject could still become ineligible prior to Angel® Catheter placement. One (1) of the six (6) enrolled (i.e. consented) subjects became ineligible prior to Angel® Catheter placement, and did not go on to start the study.
Groups:
- Angel® Catheter: All eligible subjects received an Angel® Catheter.
  The Angel® Catheter combines the functions of an inferior vena cava (IVC) filter and a multi-lumen central venous catheter (CVC). The device is designed to be placed in the inferior vena cava, via the femoral vein, for the prevention of Pulmonary Embolism (PE), and for access to the central venous system. The device is intended for short-term use (less than 30 days) and must be removed before hospital discharge.
Period: Overall Study
Arm/Group | Angel® Catheter
Started | 5 (Includes all subjects in which Angel Catheter placement was attempted.)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Angel® Catheter
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.8 (4.5)
Trauma as Primary Reason for Hospital Admission [Number; unit: participants] | 5
Baseline Venous Thromboembolism [Number; unit: participants]
  No | 5
  Yes | 0
Baseline Central Venous Catheter in Place [Number; unit: participants]
  No | 3
  Yes | 2
Subject on Mechanical Ventilation at Baseline [Number; unit: participants]
  No | 3
  Yes | 2
Subject on Vasopressors at Baseline [Number; unit: participants]
  No | 5
  Yes | 0
Subject on Dialysis at Baseline [Number; unit: participants]
  No | 5
  Yes | 0
Traumatic Brain Injury at Baseline [Number; unit: participants]
  No | 2
  Yes | 3
Subarachnoid and/or Subdural Bleeding at Baseline [Number; unit: participants]
  No | 3
  Yes | 2
Musculoskeletal Fractures at Baseline [Number; unit: participants]
  No | 1
  Yes | 4
Spinal Injury at Baseline [Number; unit: participants]
  No | 4
  Yes | 1
Respiratory Trauma or Distress at Baseline [Number; unit: participants]
  No | 1
  Yes | 4
Hepatic Trauma at Baseline [Number; unit: participants]
  No | 2
  Yes | 3
Multiple Fractures of Upper and Lower Limbs at Baseline [Number; unit: participants]
  No | 4
  Yes | 1
Spleen/Kidney Laceration at Baseline [Number; unit: participants]
  No | 3
  Yes | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Occuring for All Evaluable Subjects
Description: All Adverse Events (AEs) occurring throughout the study will be identified and characterized by seriousness, relationship to the investigational device and/or procedure, and whether un/anticipated.
Time Frame: From the time of subject enrollment through study exit (7 days post-removal or hospital discharge, whichever occurs first), for up to 37 days
Measure: Number; unit: participants
Arm/Group | Angel® Catheter
Number analyzed (Participants) | 5
participants
  Angel Catheter Related Thrombosis | 0
  Angel Catheter Related Pulmonary Embolism | 0
  Angel Catheter Related Blood Stream Infection | 0
  Angel Catheter Related Deep Vein Thrombosis (DVT) | 2
  Angel Catheter Related Major Bleeding | 0
  Angel Catheter Related Catheter Movement >2cm | 2
  Angel Catheter Related Vena Cava Perforation | 0
  Angel Catheter Related Death | 0

2. Secondary Outcome: Device Performance
Time Frame: From the time of Angel® Catheter insertion through Angel® Catheter removal, for up to 30 days
Measure: Number; unit: device malfunctions
Arm/Group | Angel® Catheter
Number analyzed (Participants) | 5
device malfunctions
  Total Number of Device Malfunctions | 2
  Device Malfunctions resulting in clinical harm | 0

ADVERSE EVENTS:
Time Frame: For all subjects in whom Angel Catheter placement was attempted, all Adverse Events were collected from the time of enrollment (i.e. consent) through study exit (i.e. after 7 days of post-removal follow-up or at hospital discharge), for up to 37 days.
Arm/Group | Angel® Catheter
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Angel® Catheter (N=5)
Deep Vein Thrombosis (Vascular disorders) | 2
Inadequate Ventilation (Respiratory, thoracic and mediastinal disorders) | 1
Perihepatic Fluid Collection (Hepatobiliary disorders) | 1
Respiratory Desaturation (Respiratory, thoracic and mediastinal disorders) | 1
Intracranial Hypertension (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Angel® Catheter (N=5)
Abnormal Chest Sounds (Respiratory, thoracic and mediastinal disorders) | 1
Constipation Related to Neurogenic Bowel (Gastrointestinal disorders) | 1
Decreased Hemoglobin (Blood and lymphatic system disorders) | 1
Decreased Hepatic Function (Hepatobiliary disorders) | 1
Decreased Phosphorus Level (Blood and lymphatic system disorders) | 1
Decreased Potassium Level (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Catheter Movement >2 cm (Surgical and medical procedures) | 2 — Because the filter is permanently attached to the catheter, filter position changes were due to movement of the entire catheter unit, not the filter. No clinical harm resulted, and the filter remained in the IVC. Reported as filter migration >2 cm.
Gastric Distention (Gastrointestinal disorders) | 1
Increased Anemia (Blood and lymphatic system disorders) | 1
Increased Platelets (Blood and lymphatic system disorders) | 1
Increased Leukocytosis (Blood and lymphatic system disorders) | 1
Pain - Abdominal (General disorders) | 2
Pain - Back (General disorders) | 1
Pain - Flank (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Vascular disorders) | 1 — PE occurred after placement of a commercial IVC filter proximal to the Angel Catheter and after Angel Catheter removal. The event was not clinically significant, and was not device or procedure related.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Tachycardia (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the small number of patients, analysis is descriptive only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No